CLINICAL TRIAL: NCT07072871
Title: The Effect of Administering the Probiotic Lactiplantibacillus Plantarum DAD-13 on Procalcitonin Levels, C-Reactive Protein, and Interleukin-6 in Sepsis Patients in the Intensive Care Unit of H. Adam Malik Hospital, Medan
Brief Title: Effect of Lactiplantibacillus Plantarum DAD-13 on Inflammatory Markers in ICU Sepsis Patients
Acronym: LactoSepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT Royal Medikalink Pharmalab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1513/KEPK/USU/2024; PT-RMP/2024 (Other: PT Royal Medicalink Pharmalab)
Record Dates: First submitted 2025-06-29; First posted 2025-07-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Sepsis; Systemic Inflammatory Response Syndrome (SIRS); Critical Illness
Keywords: Lactiplantibacillus plantarum DAD-13; Probiotics; Inflammatory markers; Procalcitonin; C-Reactive Protein; Interleukin-6; Intensive Care Unit Randomized Controlled Trial; Gut microbiota; Immune modulation
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome; Critical Illness | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, parallel-group clinical trial with two arms: probiotic and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcomes assessors were all blinded to treatment group assignments throughout the study to prevent bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Participants in this arm received placebo capsules containing maltodextrin via NGT, identical in appearance and schedule to the probiotic group (2 capsules/day for 4 days), alongside standard sepsis care.
  Interventions: Dietary Supplement: Lactiplantibacillus plantarum DAD-13; Drug: Placebo
- Dietary Supplement: Lactiplantibacillus plantarum DAD-13 (Experimental): The probiotic supplement Lactiplantibacillus plantarum DAD-13 was given in capsule form (2 capsules/day) via NGT for 4 days. Each capsule contains a standardized dose of viable bacteria formulated to modulate immune response and gut flora.
  Interventions: Dietary Supplement: Lactiplantibacillus plantarum DAD-13; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Lactiplantibacillus plantarum DAD-13 — A probiotic supplement (Vipilac®) containing Lactiplantibacillus plantarum DAD-13 administered orally via nasogastric tube, 2 capsules daily for 4 days, intended to modulate immune response and support gut microbiota in ICU sepsis patients.
  Other Names: Probiotic Group; Experimental
Drug: Placebo — Placebo capsules containing maltodextrin administered via nasogastric tube (NGT), identical in appearance and schedule to the probiotic group (2 capsules/day for 4 days), alongside standard sepsis care.
  Other Names: Control Group

SUMMARY:
This study investigated whether giving the probiotic Lactiplantibacillus plantarum DAD-13 to sepsis patients in the intensive care unit (ICU) could help reduce inflammation and improve bowel function. A total of 30 adult ICU patients with sepsis were randomly assigned to receive either the probiotic or a placebo for four days, along with standard treatment. Blood tests were performed to measure inflammatory markers, including procalcitonin (PCT), C-reactive protein (CRP), and interleukin-6 (IL-6), before and after the treatment. The study also observed defecation frequency and stool consistency. Results showed a clinical trend toward lower inflammation levels in the probiotic group and significantly better bowel function. The findings suggest that this probiotic may support immune response and gut health in sepsis patients, although more research is needed to confirm these results.

DETAILED DESCRIPTION:
This randomized controlled trial aimed to evaluate the potential benefits of the probiotic Lactiplantibacillus plantarum DAD-13 in adult ICU patients diagnosed with sepsis. The primary objective was to assess the probiotic's effect on systemic inflammation and gastrointestinal function. A total of 30 patients were randomly divided into two groups: one group received the probiotic preparation for four days in addition to standard sepsis management, while the other group received a placebo with the same treatment duration.

Inflammatory biomarkers such as procalcitonin (PCT), C-reactive protein (CRP), and interleukin-6 (IL-6) were measured before and after the intervention to evaluate immune and inflammatory responses. In addition, clinical observations were conducted on bowel movement frequency and stool consistency to assess bowel function.

The results indicated a trend toward reduced levels of inflammatory markers in the probiotic group compared to the placebo group. Moreover, patients who received the probiotic exhibited improved bowel function, including more regular defecation and better stool consistency. These findings support the hypothesis that Lactiplantibacillus plantarum DAD-13 may contribute to reducing inflammation and enhancing gut health in critically ill sepsis patients. However, due to the limited sample size, further studies are warranted to confirm the clinical significance and safety of this intervention in broader patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Diagnosed with sepsis based on clinical and laboratory criteria.
3. Admitted to ICU.
4. Receiving enteral nutrition (1500-2000 kcal/day) via nasogastric tube.
5. Able to provide or have proxy informed consent.

Exclusion Criteria:

1. History of gastrointestinal disease.
2. Immunocompromised condition (e.g., HIV, chemotherapy).
3. Presence of intravascular devices.
4. Known allergy to probiotics.
5. Concurrent participation in other clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Procalcitonin (PCT) levels in ICU sepsis patients after probiotic administration | Day 1 (T0) to Day 4 (T1) of intervention
  This outcome assesses the change in Procalcitonin (PCT) levels from baseline (day 1) to day 4 in patients with sepsis who receive Lactiplantibacillus plantarum DAD-13 or placebo. PCT is a biomarker used to evaluate the severity of systemic inflammation and response to treatment in sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Zulkarnain Zulkarnain, dr., Principal Investigator — H. Adam Malik General Hospital
Locations (1):
- H. Adam Malik General Hospital, Medan, Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-07-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT07072871/Prot_000.pdf